CLINICAL TRIAL: NCT06347172
Title: Deprescribing in Patients Living With Dementia With Caregiver and Provider Nudges
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Brown University (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Julie Lauffenburger, Associate Professor, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2024p000278; U54AG063546 (NIH)
Record Dates: First submitted 2024-03-29; First posted 2024-04-04 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Alzheimer Disease; Mild Cognitive Impairment; Dementia
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction; Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nudge internvention (Experimental): PCPs will receive an enhanced EHR alert (nudge) that triggers when a PCP opens an encounter for an eligible patient living with dementia (PLWD). The nudge will provide information about the risks of continued medication use as well as tips and tools to help providers discuss medication discontinuation with patients and care partners. Additionally, the providers will receive a brief message in their in-basket 10 days before the patient's appointment as a reminder.
  Eligible PLWD of a randomized PCP will receive the nudge intervention which includes a brief recommendation for the PLWD (and care partner, if available) via the linked patient portal prior to upcoming visits (unless explicitly opted out by the PCP) to discuss medications with the PCP at the visit and link to a general handout about medications, unless explicitly opted out by the PCP. For PLWD without a portal account, the handout will be sent to their mailing address recorded in the EHR.
  Interventions: Behavioral: Nudge Intervention

INTERVENTIONS:
Behavioral: Nudge Intervention — PCPs will receive an enhanced EHR alert (nudge) that triggers when a PCP opens an encounter for an eligible patient living with dementia (PLWD). The nudge will provide information about the risks of continued medication use as well as tips and tools to help providers discuss medication discontinuation with patients and care partners. Additionally, the providers will receive a brief message in their in-basket 10 days before the patient's appointment as a reminder.
  Eligible PLWD of a randomized PCP will receive the nudge intervention which includes a brief recommendation for the PLWD (and care partner, if available) via the linked patient portal prior to upcoming visits (unless explicitly opted out by the PCP) to discuss medications with the PCP at the visit and link to a general handout about medications, unless explicitly opted out by the PCP. For PLWD without a portal account, the handout will be sent to their mailing address recorded in the EHR.

SUMMARY:
The objectives of this study are to demonstrate the feasibility of implementing a deprescribing nudge intervention using pragmatic methods, confirm that outcomes can be feasibly measured and evaluated at scale in a subsequent embedded pragmatic clinical trial (ePCT), and explore representativeness of persons living with dementia and care partners identified.

DETAILED DESCRIPTION:
The PCP nudge will consist of: a 'pre-commitment' EHR nudge triggered when a PCP opens a patient encounter (i.e., prompt to first have a discussion and then later deprescribe) and a brief message within the in-basket prior to upcoming visits including information about their patient. The patient living with dementia (PLWD)/care partner nudge will include an electronic message delivered prior to upcoming visits (in their primary language recorded in the EHR) that includes a recommendation for the PLWD (and care partner, if available) to discuss medications with the PCP at the visit.

ELIGIBILITY:
Primary care providers will be the primary unit of identification and randomization.

Primary care providers inclusion criteria:

* Providers within Brigham and Women's Hospital primary care practices
* Having prescribed at least one of the high-risk medications of interest

Eligible patients will be identified through this providers within the health care system.

Patient inclusion criteria:

* At least 65 years of age
* Prescribed at least 90 pills of one of the high-risk medications of interest in the last 180 days in the EHR system, which most guidelines consider chronic use, and have a diagnosis of dementia in the EHR.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 250 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-10-14 (Actual); Study Completion 2025-12-15 (Actual)

PRIMARY OUTCOMES:
Composite of the percentage of eligible PCPs or their PLWD/care partners who view or click on information | On or before the primary care provider visit
  This will be the primary progression criteria for the study and measured and evaluated separately by patient and provider.

SECONDARY OUTCOMES:
Number of nudges that fire as intended: Fidelity | On the primary care provider visit
  Number of nudges that fired as intended
Discontinuation or prescribed reduction in medication | Within 60 days after the primary care provider visit
  Discontinuation or prescribed reduction in dose of at least one high-risk medication of interest within 60 days after the visit.

CONTACTS AND LOCATIONS:
Overall Officials: Julie Lauffenburger, PharmD, PhD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Mass General Brigham, Boston, Massachusetts, United States